CLINICAL TRIAL: NCT01971216
Title: Mother-infant Signalling During Breastfeeding: A Randomised Trial Investigating the Effects of a Relaxation Intervention in Breastfeeding Mothers on Breast Milk Production, Breast Milk Cortisol and Infant Behaviour and Growth.
Brief Title: Mother-infant Signalling During Breastfeeding
Acronym: MOMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 13NT05
Record Dates: First submitted 2013-10-23; First posted 2013-10-29 (Estimated); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Breastfeeding Women
Keywords: Breastfeeding, relaxation, anxiety, infant growth
MeSH Terms: conditions — Breast Feeding; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Breastfeeding mothers who are not randomised to relaxation intervention
- Relaxation (Experimental): Breastfeeding mothers randomised to use relaxation tape at 2 weeks post-partum
  Interventions: Behavioral: Relaxation

INTERVENTIONS:
Behavioral: Relaxation
  Other Names: Relaxation tape - audio tape with visual imagery and relaxation exercises
  Arms: Relaxation

SUMMARY:
Primary hypotheses

1. The use of a relaxation tape by breastfeeding mothers that will be given starting at week 2 postpartum, will result in : i) reduced maternal stress and anxiety ii) the production of a higher volume of breast milk iii) lower milk cortisol concentrations iv) favourable effects on infant behaviour (less crying, more sleeping) v) higher milk intake by the infant vi) more optimal growth, specifically higher lean mass and lower fat mass (body composition)

Secondary hypotheses (i) Infant temperament/behaviour and gender influence milk and energy intake and hence early growth and body composition (ii) Non-nutrient factors in breast milk (hormones including ghrelin and leptin) influence infant behaviour and feeding patterns and hence infant growth and body composition.

ELIGIBILITY:
Inclusion Criteria:

Primiparous mother with singleton pregnancy Infant is singleton and born at term (37-42 week of gestation) Infant birth weight of >2500 g (5,5 pounds or 5 pounds and 8,2 ounces) Mother and infant are generally healthy (free of serious illness that can affect breastfeeding or nursing infant, or energy balance of the infant).

No current or recent involvement in other research studies that could potentially affect any of outcome measures.

Mother speaks and understands either English only or English and Malay (some questionnaires are in English)

Exclusion Criteria:

Mother or baby has a major illness that affects nursing or breastfeeding, or affects energy balance of the infant.

Mother smokes Mothers who do not exclusively breastfeed their infant

-

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2015-03 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Maternal stress and anxiety | Baselibne to 12 weeks
  Maternal stress and anxiety assessed using the Cohen's Perceived Stress Scale (PSS) and Beck Anxiety Inventory (BAI) respectively (change in score from baseline to end-point at 12 weeks)
Breast milk volume at 12 weeks assessed non-invasively using stable isotope techniques | 12 weeks
  Breast milk volume at 12 weeks assessed non-invasively using stable isotope techniques
Breast milk cortisol concentrations at 12 weeks | 12 weeks
Infant behaviour measured using a 3-day diary at 12 weeks | 12 weeks
Infant weight and body composition measured using stable isotopes at 12 weeks | 12 weeks
Physiological changes (maternal saliva cortisol, breast milk cortisol and milk volume) before and after physiological-mini test in intervention group at 2,6 and 12 weeks. | 2,6,12 weeks

SECONDARY OUTCOMES:
Non-nutrient factors in breast milk - leptin and ghrelin | 2,6,12 weeks
Macronutrient composition of breast milk (fat and protein) | 2,6,12 weeks

OTHER OUTCOMES:
Infant temperament measured using the Rothbart questionnaire | 12 weeks
Infant appetite assessed using the BEBQ | 2,6,12 weeks
Maternal depression assessed using Edinburgh Postnatal Depression Scale (EPDS) | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mary Fewtrell, MD, Principal Investigator — UCL Institute of Child Health, London
Locations (1):
- Faculty of Medicine and Health Science, Universiti Putra Malaysia (UPM)., Kuala Lumpur, Malaysia

REFERENCES:
- [Derived] Mohd Shukri NH, Wells J, Eaton S, Mukhtar F, Petelin A, Jenko-Praznikar Z, Fewtrell M. Randomized controlled trial investigating the effects of a breastfeeding relaxation intervention on maternal psychological state, breast milk outcomes, and infant behavior and growth. Am J Clin Nutr. 2019 Jul 1;110(1):121-130. doi: 10.1093/ajcn/nqz033. PMID 31161202
- [Derived] Shukri NHM, Wells J, Mukhtar F, Lee MHS, Fewtrell M. Study protocol: An investigation of mother-infant signalling during breastfeeding using a randomised trial to test the effectiveness of breastfeeding relaxation therapy on maternal psychological state, breast milk production and infant behaviour and growth. Int Breastfeed J. 2017 Jul 14;12:33. doi: 10.1186/s13006-017-0124-y. eCollection 2017. PMID 28725257